CLINICAL TRIAL: NCT04368013
Title: Host-pathogen Interactions, Immune Response, and Clinical Prognosis at COVID-19 - the CoVUm Trial
Acronym: CoVUm
Status: Active, not recruiting | Type: Observational
Sponsor: Johan Normark (Other)
Collaborators: Umeå University (Other); Region Västerbotten (Other Government); Örebro University, Sweden (Other); Värmland County Council, Sweden (Other Government); Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor-Investigator, Johan Normark, Associate professor, Umeå University
Organization: Umeå University (Other)
Other Study IDs: CoVUm
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, Stool, Urine, nasopharynx swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: The difference from the standard of care is extended sample collection and study related procedures during the study.
  Interventions: Procedure: Extended sampling and procedures

INTERVENTIONS:
Procedure: Extended sampling and procedures — The study patients will give additional blood samples and also urine and faeces samples. Spirometry and additional biometric controls will be performed regularly. Necrobiopsies of various organs from deceased patients will be secured and stored for immunohistological and virological analysis.

SUMMARY:
The project aims to clarify how immunity to SARS-CoV2 develops in humans and to investigate the possibility of finding patients with a particularly effective, neutralizing antibody response for future treatment. The project also aims to detail the virus's damage mechanisms in tissue.

DETAILED DESCRIPTION:
There is currently a mounting body of evidence regarding the pathogenesis of COVID-19 caused by SARS-CoV2. By gaining more knowledge about the mechanisms in the development of viral pneumonia and the influence of other organ systems at SARS-CoV2, we believe that in the future it is better to be able to identify precisely those persons who are at risk of serious illness. To this we will gain knowledge of how humans develops immunity to the virus and also how human epigenetic (acquired) ability to activate inflammatory genetic systems can limit the harmful effects of the virus. Thus, patients who have had mild or no symptoms are just as interesting from a study point of view as those who have had severe symptoms. Hopefully, such understanding can also contribute to other opportunities for targeted treatment (by identifying patients who can mount effective inborn and adaptive host defenses) in order to prevent severe disease and death in pandemic corona infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 15-100 years with SARS-CoV2 or influenza
* Patients admitted for COVID-19 or Influenza-caused pneumonia/ pneumonitis at the Departments of Infectious Diseases or ICU, Umeå University Hospital, Örebro hospital, Karlstad hospital and Västerås hospital
* Patients with COVID-19 who are treated in outpatient care at the infectious Diseases Clinic, Umeå University Hospital, Sweden
* Patients who give written informed consent to participate in the study for the entire follow- up period of 5 years.

Exclusion Criteria:

* Age less than 15 years

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A mixed population of individuals suffering from Covid-19 or influenza
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Mortality | Five years after study start
  Deceased or alive at five year follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Incectious Diseases Clinic, Umeå, Västerbotten County
  - Karlstad hospital, Karlstad
  - Örebro university hospital, Örebro
  - Västerås hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staessen JA, Wendt R, Yu YL, Kalbitz S, Thijs L, Siwy J, Raad J, Metzger J, Neuhaus B, Papkalla A, von der Leyen H, Mebazaa A, Dudoignon E, Spasovski G, Milenkova M, Canevska-Taneska A, Salgueira Lazo M, Psichogiou M, Rajzer MW, Fulawka L, Dzitkowska-Zabielska M, Weiss G, Feldt T, Stegemann M, Normark J, Zoufaly A, Schmiedel S, Seilmaier M, Rumpf B, Banasik M, Krajewska M, Catanese L, Rupprecht HD, Czerwienska B, Peters B, Nilsson A, Rothfuss K, Lubbert C, Mischak H, Beige J; CRIT-CoV-U investigators. Predictive performance and clinical application of COV50, a urinary proteomic biomarker in early COVID-19 infection: a prospective multicentre cohort study. Lancet Digit Health. 2022 Oct;4(10):e727-e737. doi: 10.1016/S2589-7500(22)00150-9. Epub 2022 Aug 31. PMID 36057526
- [Result] Schagatay F, Diamant K, Liden M, Edin A, Athlin S, Hultgren O, Ahlm C, Forsell MNE, Savilampi J, Normark J, Lange A, Cajander S. Serum concentration of extracellular cold-inducible RNA-binding protein is associated with respiratory failure in COVID-19. Front Immunol. 2022 Jul 29;13:945603. doi: 10.3389/fimmu.2022.945603. eCollection 2022. PMID 35967397
- [Result] Zhou S, Butler-Laporte G, Nakanishi T, Morrison DR, Afilalo J, Afilalo M, Laurent L, Pietzner M, Kerrison N, Zhao K, Brunet-Ratnasingham E, Henry D, Kimchi N, Afrasiabi Z, Rezk N, Bouab M, Petitjean L, Guzman C, Xue X, Tselios C, Vulesevic B, Adeleye O, Abdullah T, Almamlouk N, Chen Y, Chasse M, Durand M, Paterson C, Normark J, Frithiof R, Lipcsey M, Hultstrom M, Greenwood CMT, Zeberg H, Langenberg C, Thysell E, Pollak M, Mooser V, Forgetta V, Kaufmann DE, Richards JB. A Neanderthal OAS1 isoform protects individuals of European ancestry against COVID-19 susceptibility and severity. Nat Med. 2021 Apr;27(4):659-667. doi: 10.1038/s41591-021-01281-1. Epub 2021 Feb 25. PMID 33633408
- [Result] Bystrom JW, Vikstrom L, Rosendal E, Groning R, Gwon YD, Nilsson E, Sharma A, Espaillat A, Hanke L, McInerney G, Puhar A, Cava F, Karlsson Hedestam GB, Thunberg T, Monsen T, Elgh F, Evander M, Johansson AF, Overby AK, Ahlm C, Normark J, Forsell MN. At-home sampling to meet geographical challenges for serological assessment of SARS-CoV-2 exposure in a rural region of northern Sweden, March to May 2021: a retrospective cohort study. Euro Surveill. 2023 Mar;28(13):2200432. doi: 10.2807/1560-7917.ES.2023.28.13.2200432. PMID 36995373
- [Result] Bjorsell T, Sundh J, Lange A, Ahlm C, Forsell MNE, Tevell S, Blomberg A, Edin A, Normark J, Cajander S. Risk factors for impaired respiratory function post COVID-19: A prospective cohort study of nonhospitalized and hospitalized patients. J Intern Med. 2023 May;293(5):600-614. doi: 10.1111/joim.13614. Epub 2023 Feb 23. PMID 36815689
- [Result] Ahmad I, Edin A, Granvik C, Kumm Persson L, Tevell S, Mansson E, Magnuson A, Marklund I, Persson IL, Kauppi A, Ahlm C, Forsell MNE, Sundh J, Lange A, Cajander S, Normark J. High prevalence of persistent symptoms and reduced health-related quality of life 6 months after COVID-19. Front Public Health. 2023 Feb 2;11:1104267. doi: 10.3389/fpubh.2023.1104267. eCollection 2023. PMID 36817925